CLINICAL TRIAL: NCT06262789
Title: RAT-HEMATO : Return to Work After Malignant Hemopathy
Acronym: RAT-HEMATO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 49RC23_0011
Record Dates: First submitted 2024-01-26; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm with "return-to-work after cancer" consultation (Experimental)
  Interventions: Other: "Return-to-work after cancer" consultation
- Standard arm without with "return-to-work after cancer" consultation (No Intervention): Patient are treated according to usual care, according to local practice.

INTERVENTIONS:
Other: "Return-to-work after cancer" consultation — The "return-to-work after cancer" consultation is carried out by a specialist in occupational pathology, who may be assisted by a psychologist and/or a nurse and/or a social worker, depending on the patient's personal situation. During this consultation, the team assesses the patient's medical situation, social situation and psychological situation. This consultation lasts approximatively 1 hour and aims to guide the patient in the different stages of return to work, to identify obstacles and apprehensions about return to work, to assess the patient's functional capacities and motivations, to provide information on the legislation, actors and tools for employment maintenance and to discuss possible adjustments of the work situation. The consultation provides a response to potential or encountered problems, directs the patient towards the actors and tools adapted to his/her situation.
  Arms: Experimental arm with "return-to-work after cancer" consultation

SUMMARY:
Return to work (RTW) of patients after cancer treatment has been a topic of growing interest for the past two decades. Advances in cancer care have led to better patient survival, with some cancers considered as chronic or even cured diseases. The return of patients to their "pre-cancer life" can thus become an objective. Indeed, RTW after cancer is associated with improved quality of life for patients in several studies (improved financial status, improved social contacts, return of functional abilities and improved self-esteem). However, many difficulties can interfere with RTW. Many factors have been identified: disease, treatment, patient and occupational factors. The feeling of "return-to-work self-efficacy" is one of the main psychological determinants and its interest has been recently demonstrated in oncology. It corresponds to a cognitive mechanism based on expectations and/or beliefs of an individual about being able to carry out the actions required to achieve a goal, in this case RTW. The majority of studies on RTW concerns solid cancer and are retrospective. Very few studies have focused on hematological malignancies, whose prognosis was, until recently, worse. Moreover, very few interventional studies exist. There is therefore a significant need for prospective studies with appropriate methodological tools to reliably assess the benefit of interventional measures on RTW. The investigators propose to conduct a prospective, comparative, randomized, multicenter study evaluating the impact of an early RTW-consultation in patients who have been treated for a hematological malignancy. The investigators hypothesize that this consultation will improve patients' RTW rates and RTW quality.

ELIGIBILITY:
Inclusion Criteria :

* Patient with hematological malignancy controlled after treatment
* Induction/consolidation chemotherapy completed (excluding maintenance therapy)
* Patient aged 18 to 55
* Patient having worked at least 6 months in the 2 years before diagnosis of hematological malignancy
* Patient who has not yet returned to work since diagnosis of hematological malignancy
* Signed informed consent form

Exclusion Criteria:

* Patient choosing not to return to work
* Patient not affiliated to a social security system
* Patient with legal guardian or legal trustee
* Patient not understanding French
* Patient with severe cognitive impairment at diagnosis, incompatible with the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 264 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Return-to-work rate at 1 year (percentage) | 12 months
  The return-to-work rate at 1 year is used to assess the impact of an early "Return-to-work" after cancer consultation for patients with hematological malignancies. It is defined as the percentage of patients having returned to work, including part-time work, 1 year after the inclusion visit.

SECONDARY OUTCOMES:
Cumulative incidence of return-to-work at 1 year | 12 months
  It is measured by the cumulative incidence rate of return-to-work at 1 year
Change or not of the professional situation in the 2 arms | 12 months
  It is defined as the rate of patients with a change of their professional situation since the diagnosis. The changes of professional situation include: employment yes/no, full-time/part-time work, adaptation of work station yes/non, change of profession compared to before diagnosis.
Factors influencing return to work | 12 months
  The factors investigated are type of hematological malignancy, sex, type of profession, presence of anxio-depressive disorders
Quality of life (SF-12 score) evolution | Baseline, 3 months, 6 months and 12 months
  The 12-Item Short Form Survey (SF-12) is one of the most widely used tools in oncology to assess health-related quality of life. It is a general health questionnaire that measures physical and mental health. It consists of 12 questions split into 8 different dimensions: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional and mental health. Results are expressed in terms of two meta-scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). PCS and MCS scores range from 0 to 100, with higher scores indicating better physical and mental health functioning, respectively.
  We will evaluate SF-12 evolution between Baseline visit and each other visits.
Anxiety and depression (HAD scale) evolution | Baseline , 3 months, 6 months and 12 months
  Hospital Anxiety and Depression Scale (HAD scale) is one the most widely tools used in oncology to assess patient anxiety and depression. It consists of 14 questions rated form 0 to 3: 7 questions relate to anxiety (total A) and 7 to depression (total D), giving two scores (maximum score for each = 21). Scores between 0 et 7 correspond to an absence of anxiety or depression, scores between 8 and 10 are considered as doubtful, and scores 11 and above correspond to depression or anxiety.
  We will evaluate HAD scale evolution between Baseline visit and each other visits.
Return-to-work self-efficacy (RTW-SE-11 scale) evolution | Baseline, 3 months, 6 months and 12 months
  The Return-to-Work Self-Efficacy Scale - 11 items (RTW-SE-11) is an 11-item questionnaire measuring an individual's confidence in his or her ability to return to work. It integrates beliefs in the patient's abilities to support the physical, cognitive, emotional, relational and professional aspects of the work environment that have been identified as strong predictors of RTW following a cancer diagnosis. The final score ranges between 1 and 6, with a higher score indicating higher self-efficacy.
  We will evaluate RTW-SE-11 scale evolution between Baseline visit and each other visits.
Self-assessment of the benefit of the "return-to-work after cancer" consultation | 3 months and 6 months
  Patients assess the benefit of the "return-to-work after cancer" consultation using a questionnaire specially designed for the study, composed of Likert-scale questions. For each question, score ranges from 1 to 5. Higher scores indicate higher satisfaction.
  We will evaluate RTW-SE-11 scale evolution between 3 months visit and 6 months visit (only for patients randomized in intervention arm).

CONTACTS AND LOCATIONS:
Overall Officials: Jérome PAILLASSA, MD, Principal Investigator — University Hospital, Angers
Locations (7):
- France (7):
  - Angers University hospital, Angers
  - Brest University Hospital, Morvan Site, Brest
  - Caen University hospital, Caen
  - Rennes University Hospital, Pontchaillou site, Rennes
  - Centre Henri Becquerel, Rouen
  - Rouen University Hospital, Rouen
  - Tours University Hospital, Bretonneau Site, Tours

IPD SHARING:
Plan to Share IPD: No